CLINICAL TRIAL: NCT05196425
Title: Expression of PARP-1 in Optic Neuritis of Multiple Sclerosis Patients
Brief Title: Expression of PARP-1 in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Lecturer of ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-05-12
Record Dates: First submitted 2021-12-07; First posted 2022-01-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: Optic neuritis-Multiple sclerosis-PARP-1
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other)
  Interventions: Genetic: Blood sampling
- MS with optic neuritis (Active Comparator)
  Interventions: Genetic: Blood sampling
- Ms without optic neuritis (Active Comparator)
  Interventions: Genetic: Blood sampling

INTERVENTIONS:
Genetic: Blood sampling — Blood sample for detection of PARP-1 gene and correlate to changes of the optic disc, RNFL and GCC layers of the retina of MS patients

SUMMARY:
This study will explore the expression of PARP-1 in optic neuritis of multiple sclerosis patients.

The data will be collected from Sohag University hospital in the period from the start of August 2021 to the end of December 2021.

The study protocol will be approved by the Scientific Research Ethical Committee, Faculty of Medicine, Sohag University.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis with or without optic neuritis Multiple sclerosis will be diagnosed according to the McDonald criteria

Exclusion Criteria:

* • Isolated optic neuritis.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
measure PARP-1 mRNA | 2 weeks
  measure PARP-1 mRNA

SECONDARY OUTCOMES:
Optic nerve, RNFL and GCC layer affection by MS | 2 weeks
  Optic nerve Retinal nerve fibre layer (RNFL) in um
  ) and Ganglion cell complex (GCC) layer affection in um by MS in correlation to PARP-1 mRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Elshimaa A.Mateen, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided